CLINICAL TRIAL: NCT04373629
Title: Neural Mechanisms of Perceptual Abnormalities and Their Malleability in Body Dysmorphic Disorder
Brief Title: Perceptual Abnormalities and Their Malleability in BDD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre for Addiction and Mental Health (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH); University of Alabama at Birmingham (Other); University of Toronto (Other)
Responsible Party: Principal Investigator, Jamie D. Feusner, Professor of Psychiatry, Centre for Addiction and Mental Health
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: R01MH121520-01A1 (NIH); R01MH121520 (NIH)
Record Dates: First submitted 2020-04-24; First posted 2020-05-04 (Actual); Last update posted 2025-11-14 (Actual); Status verified 2025-11

CONDITIONS: Body Dysmorphic Disorder
MeSH Terms: conditions — Body Dysmorphic Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- attention modulation (Experimental)
  Interventions: Behavioral: attentional modulation
- perceptual modulation (Experimental)
  Interventions: Other: perceptual modulation
- naturalistic viewing (Experimental)
  Interventions: Other: naturalistic viewing

INTERVENTIONS:
Behavioral: attentional modulation — Attentional instructions when viewing faces will be given
  Arms: attention modulation
Other: perceptual modulation — Faces will be presented of varying durations
  Arms: perceptual modulation
Other: naturalistic viewing — Faces will be viewed without specific instructions
  Arms: naturalistic viewing

SUMMARY:
A core symptom of body dysmorphic disorder (BDD) is perceptual distortions for appearance, which contributes to poor insight and delusionality, limits engagement in treatment, and puts individuals at risk for relapse. Results from this study will provide a comprehensive mechanistic model of brain, behavioral, and emotional contributors to abnormal perceptual processing, as well as how malleable it is with visual modulation techniques. This will lay the groundwork for next-step translational perceptual retraining approaches.

DETAILED DESCRIPTION:
Individuals with body dysmorphic disorder (BDD) misperceive specific aspects of one's own appearance to be conspicuously flawed or defective, despite these being unnoticeable or appearing minuscule to others. With convictions of disfigurement and ugliness, individuals with BDD typically have poor insight or delusional beliefs, obsessive thoughts and compulsive behaviors, anxiety, and depression. These result in significant difficulties in functioning, depression, suicide attempts (25%), and psychiatric hospitalization (50%). Despite this, relatively few studies of the neurobiology, and few treatment studies, have been conducted. This underscores a critical need for research to identify novel targets for intervention based on a comprehensive understanding of the pathophysiological mechanisms. Neuropsychological, behavioral, and neurobiological research by investigators have uncovered mechanisms that may contribute to perceptual distortions, including prominent abnormalities in visual processing systems. These have contributed to a model of diminished global/holistic processing and enhanced local/detailed processing, attributed to "bottom-up" and "top-down" disturbances in perception. Using psychophysical experiments and novel visual modulation techniques, investigators have probed the brain's visual systems responsible for global and local processing and found early evidence that they may be modifiable in BDD. These techniques include a "top-down" attentional modulation and a "bottom-up" perceptual modulation strategy. Abnormal eye gaze and emotional arousal when viewing faces may further contribute to abnormal perception. Whether these brain and behavior abnormalities are directly linked to abnormal perception remains to be understood. Accordingly, this study will determine a) if abnormalities in neural activation and connectivity in BDD when viewing one's own appearance are directly associated with abnormalities in perceptual functioning; and b) if changes in neural activation and connectivity from these visual modulation strategies are linked to changes in perceptual functioning, thus representing potential biomarkers. Investigators will also determine how attentional systems, eye gaze behaviors and emotional arousal interact with brain functioning in visual systems, and with global and local perceptual functioning. Investigators will enroll participants with BDD, with subclinical BDD, and healthy controls who will undergo functional magnetic resonance imaging while viewing photographs of own, and others' faces. Investigators will obtain measures of global and local visual processing, emotional arousal while participants view own face, and eye gaze behaviors using eye tracking. To understand the malleability of global/local perception, and the neural mechanisms of these changes, investigators will determine whether repeated visual modulation using top-down and bottom-up strategies results in alterations of perceptual functioning and brain activity/connectivity, and relationships between them. Results will provide a comprehensive mechanistic model of abnormal visual information processing underlying the core symptom domain of misperceptions of appearance. This will lay the groundwork for next-step translational approaches.

ELIGIBILITY:
Inclusion Criteria:

Body dysmorphic disorder: Inclusion:

* males or females
* ages 18-40
* meet Diagnostic and Statistical Manual-5 (DSM-5) criteria for Body Dysmorphic Disorder
* have a Body Dysmorphic Disorder version of the Yale-Brown Obsessive-Compulsive Disorder Scale (BDD-YBOCS) score of ≥20
* primary appearance concerns of the face or head area
* medication naïve or medication free for at least 8 weeks prior to enrollment

Inclusion Criteria:

Subclinical body dysmorphic disorder: Inclusion:

* males or females
* ages 18-40
* have a score on the Dysmorphic Concern Questionnaire of ≥8 [1 standard deviation (STD) above population norms] - primary appearance concerns of the face or head area
* medication naïve or medication free for at least 8 weeks prior to enrollment

Inclusion Criteria:

Healthy controls: Inclusion

* Healthy males and females from any racial or ethnic background - ages 18-40
* have a score on the Dysmorphic Concern Questionnaire of <8

Exclusion Criteria:

Body dysmorphic disorder: Exclusion

* concurrent major Axis I disorders including substance use disorders, aside from anxiety disorders or depressive disorders, as these comorbidities are very common and the sample would otherwise be non-representative; however BDD must be the primary diagnosis.
* lifetime: bipolar disorder or psychotic disorder.
* psychotropic medications, aside from a short half-life sedative/hypnotic for insomnia, or a short half-life benzodiazepine as needed for anxiety but not exceeding a frequency of 3 doses in one week and not to be taken on the days of the training or MRI scan
* current cognitive-behavioral therapy

Exclusion:

Subclinical body dysmorphic disorder: Exclusion

* meet full DSM-5 criteria for Body Dysmorphic Disorder
* current Axis I disorders including substance use disorders
* lifetime: bipolar disorder or psychotic disorder
* psychotropic medications, aside from a short half-life sedative/hypnotic for insomnia, or a short half-life benzodiazepine as needed for anxiety but not exceeding a frequency of 3 doses in one week and not to be taken on the days of the training or MRI scan
* current cognitive-behavioral therapy

Exclusion Criteria:

Healthy Controls: Exclusion

* Any current Axis I disorder
* lifetime: bipolar disorder or psychotic disorder
* Psychiatric medication

Exclusion Criteria:

All participants: Exclusion

* Neurological disorder
* Pregnancy
* Current major medical disorders that may affect cerebral metabolism such as diabetes or thyroid disorders - Current risk of suicide with a plan and intent
* Ferromagnetic metal implantations or devices (electronic implants or devices, infusion pumps, aneurysm clips, metal fragments or foreign bodies, metal prostheses, joints, rods or plates)
* Visual acuity worse than 20/35 for each eye as determined by Snellen close vision acuity chart (vision will be tested with corrective lenses if participant uses them).

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 146 (Estimated)
Dates: Start 2020-12-01 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Face inversion effect | Baseline
  In a force-choice recognition task, participants will view sets of upright target faces followed by 2 upright selection faces, and sets of inverted target faces followed by 2 inverted selection faces. Participants will be instructed to select one of the two faces that is the same as the target face, as quickly and as accurately as possible. The dependent variable is the difference in response times for upright vs. inverted faces.
Brain connectivity and activation in the dorsal and ventral visual stream | Baseline
  Investigators will obtain functional magnetic resonance imaging (fMRI) data while participants view photographs of one's face. After preprocessing and analysis investigators will be able to determine: a) baseline associations between brain activity and connectivity and global/ local processing (face inversion effect), and b) associations between changes in brain activity and connectivity with changes in global/local processing (face inversion effect)
Eye gaze behavior | Baseline
  Investigators will use eye-tracking for behavioral assessments related to viewing photos of one's face. The primary dependent variable will be mean fixation duration, defined as the mean time that eye gaze is limited to one area (using k-means clustering) across the total viewing duration. We will use an eye-tracker camera to collect data while individuals view photos of one's face. Each face will be 3.5 sec.
Emotional valence | Baseline
  Investigators will use automated facial emotional recognition software to calculate valence based on the activity of specific facial landmarks automatically read from video capture of participants while viewing one's own face. The data will be collected simultaneously with the eye-tracking data collection while viewing own faces. The dependent variable of emotional is calculated as the mean, across the entire face viewing, of the intensity of positive emotional expressions minus the intensity of the negative expression with the highest intensity.
Change in face inversion effect | Within a week after baseline
  In a force-choice recognition task, participants will view sets of upright target faces
Change in brain connectivity and activation in the dorsal and ventral visual stream | Within a week after baseline
  Investigators will obtain functional magnetic resonance imaging (fMRI) data while participants view photographs of one's own face. After preprocessing and analysis investigators will be able to determine: a) baseline associations between brain activity and connectivity and global/ local processing (face inversion effect), and b) associations between changes in brain activity and connectivity with changes in global/local processing (face inversion effect)
Change in eye gaze behavior | Within a week after baseline
  Investigators will use eye-tracking for behavioral assessments related to viewing photos of one's face. The primary dependent variable will be mean fixation duration, defined as the mean time that eye gaze is limited to one area (using k-means clustering) across the total viewing duration. Investigators will use an eye-tracker camera to collect data while individuals view photos of one's own face. Each face will be 3.5 sec.
Change in emotional valence | Within a week after baseline
  Investigators will use automated facial emotional recognition software to calculate valence based on the activity of specific facial landmarks automatically read from video capture of participants while viewing one's own face. The data will be collected simultaneously with the eye-tracking data collection while viewing own faces. The dependent variable of emotional is calculated as the mean, across the entire face viewing, of the intensity of positive emotional expressions minus the intensity of the negative expression with the highest intensity.

SECONDARY OUTCOMES:
The body dysmorphic version of the Yale-Brown Obsessive-Compulsive Scale 0-48 values higher score= worse outcome | Baseline
  This is the most widely used scale to measure BDD symptom severity cross-sectionally, and as a measure of symptom change in treatment studies. It is a clinician-rated scale that consists of 12 items assessing appearance-related obsessions, compulsive behaviors, insight, and avoidance.
The Brown Assessment of Beliefs Scale 0-24 values higher score= worse outcome | Baseline
  This clinician-rated scale assesses insight and delusionality related to specific beliefs. It consists of six items that probe one's convictions about their beliefs, if others' agree with their beliefs, attempts to disprove their beliefs, and if their beliefs have psychological or psychiatric causes.
Body Image States Scale 1-9 values higher the score= better outcome | Baseline
  This scale consists of six items to assess domains of current body experiences
Change in the body dysmorphic version of the Yale-Brown Obsessive- Compulsive Scale 0-48 values higher score= worse outcome | 7-10 days after baseline
  This is the most widely used scale to measure BDD symptom severity cross-sectionally, and as a measure of symptom change in treatment studies. It is a clinician-rated scale that consists of 12 items assessing appearance-related obsessions, compulsive behaviors, insight, and avoidance.
Change in the Brown Assessment of Beliefs Scale 0-24 values higher score= worse outcome | 7-10 days after baseline
  This clinician-rated scale assesses insight and delusionality related to specific beliefs. It consists of six items that probe one's convictions about their beliefs, if others' agree with their beliefs, attempts to disprove their beliefs, and if their beliefs have psychological or psychiatric causes.
Change in the Body Image States Scale 1-9 values higher the score= better outcome | 7-10 days after baseline
  This scale consists of six items to assess domains of current body experiences

CONTACTS AND LOCATIONS:
Overall Officials: Jamie D Feusner, M.D., Principal Investigator — Centre for Addiction and Mental Health
Locations (1):
- Centre for Addiction and Mental Health, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No